CLINICAL TRIAL: NCT06682884
Title: Phase II, Open-label, Single-arm, Prospective, Multi-center Study to Evaluate the Efficacy and Safety of Lorlatinib as Neoadjuvant Treatment in Surgically Resectable Stage IB-IIIB ALK-rearranged Non-Small Cell Lung Cancer (NEOLORA)
Brief Title: Lorlatinib as Neoadjuvant Treatment in Stage IB-IIIB ALK-rearranged Non-Small Cell Lung Cancer
Acronym: NEOLORA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: Hunan Cancer Hospital (Other); Liaoning Cancer Hospital & Institute (Other); Air Force Military Medical University, China (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Yang Fan, MD, Professor of Thoracic Surgery, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024PHD022-002
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Neoadjuvant Non-Small Cell Lung Cancer
Keywords: NSCLC; Neoadjuvant; ALK-rearranged; Lorlatinib
MeSH Terms: interventions — lorlatinib

STUDY DESIGN:
Intervention Model Description: Lorlatinib as Neoadjuvant Treatment in Stage IB-IIIB ALK-rearranged Non-Small Cell Lung Cancer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lorlatinib as Neoadjuvant Treatment (Experimental): These patients will receive lorlatinib neoadjuvant therapy for 6-8 weeks (determined by clinicians' decision based on clinical practice) and then underwent surgery
  Interventions: Drug: Lorlatinib 100 mg

INTERVENTIONS:
Drug: Lorlatinib 100 mg — Eligible patients will be registered to receive oral lorlatinib 100mg qd for 6-8 weeks each during the neoadjuvant therapy phase
  Other Names: third generation ALK- TKI

SUMMARY:
This project was designed To explore the pathological complete response (pCR) of lorlatinib as neoadjuvant treatment. Twenty-five patients will be involved in this study.

These patients will receive lorlatinib neoadjuvant therapy for 6-8 weeks (determined by clinicians' decision based on clinical practice) and then underwent surgery.

Previous small-sample clinical studies on ALK inhibitors as neoadjuvant therapy in resectable NSCLC have shown promising outcomes including MPR and pCR, supporting the potential of ALK TKIs in this setting.

DETAILED DESCRIPTION:
Lung cancer remains the foremost cause of cancer-related deaths worldwide, with non-small cell lung cancer (NSCLC) constituting approximately 80% of all lung cancer cases. 1Despite advancements, the prognosis for NSCLC patients, particularly those ineligible for surgical resection at diagnosis, is dismal, with median 5-year overall survival (OS) rates between 36% and 60%. 2Currently, neoadjuvant (preoperative) platinum-based doublet chemotherapy regimens represent the standard care for resectable stage II or III NSCLC with oncogenic driver mutations. However, the marginal improvement in long-term survival underscores the critical need for more effective treatment strategies.3 The discovery of driver mutations in NSCLC has revolutionized treatment approaches, with alterations in the anaplastic lymphoma kinase (ALK) gene being one of the significant breakthroughs. ALK rearrangements are identified in 3%-7% of NSCLC cases, guiding the development of targeted therapies. ALK inhibitors, including crizotinib, ceritinib, alectinib, brigatinib, and notably lorlatinib, have significantly impacted the treatment landscape of ALK-positive NSCLC by offering substantial improvements in survival and disease control.

Lorlatinib, a potent third-generation ALK inhibitor, is distinguished by its efficacy against a wide spectrum of ALK mutations, including those conferring resistance to earlier generations of ALK inhibitors. Its ability to cross the blood-brain barrier presents an added advantage for controlling central nervous system (CNS) metastases, a frequent challenge in NSCLC management. This profile, along with encouraging outcomes from phase I and II trials demonstrating lorlatinib's robust antitumor activity in patients who have progressed on previous ALK TKI therapies, underscores its potential as a transformative neoadjuvant therapy option. 4-6 The advent of targeted therapies has markedly shifted the paradigm in the treatment of non-small cell lung cancer (NSCLC), particularly for patients with specific genetic alterations such as ALK rearrangements. A small retrospective study of the first-generation ALK-TKI crizotinib in the neoadjuvant setting included 11 ALK-positive, N2 NSCLC patients who received oral crizotinib (250mg twice daily) for a median duration of 30 days (range 28-120 days). This study demonstrated a 91.0% R0 resection rate with 18.2% (2 cases) achieving pathological complete response post-treatment.7 The SAKULA study, a phase II multicenter single-arm trial, assessed the efficacy and safety of the second-generation ALK-TKI ceritinib in resectable ALK-positive NSCLC. The study enrolled 7 cases all at stage IIIA (N2), and treated with oral ceritinib (750mg twice daily) as neoadjuvant therapy. The primary endpoint of major pathological response (MPR) was 57% (95% CI: 18-90), with 2 cases achieving complete remission (29%). 8NAUTIKA1, a phase II trial, investigated the efficacy of alectinib as neoadjuvant therapy for 8 weeks in patients with resectable stage II, IIIA, and IIIB NSCLC, followed by surgery, 4 cycles of adjuvant chemotherapy, and 2 years of alectinib adjuvant treatment. Among 9 patients, 6 achieved a major pathological response (MPR), resulting in an MPR rate of 66.7% (95%CI, 29.9%-92.5%), with a pathological complete response (pCR) rate of 33.3%. Eight patients underwent R0 resection. 9These results indicate the feasibility and potential efficacy of ALK-TKIs in improving surgical outcomes and reducing the tumor burden before surgery, making it a promising neoadjuvant treatment option for this patient population.

This study seeks to assess the feasibility of lorlatinib as neoadjuvant therapy for patients with resectable, stage IB-IIIB ALK+ lung adenocarcinoma. Given lorlatinib's advanced efficacy in targeting ALK-positive tumors, including its activity against resistant mutations and its proficiency in managing CNS metastases,This study aims to evaluate the efficacy and safety of lorlatinib as neoadjuvant therapy in patients, focusing on improvements in pathological response, surgical outcomes, prolonged survival, and safety/tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Imaging confirmed, resectable stage IB, II, IIIA or selected IIIB (including T4N2，per AJCC 8th edition)
* Histologically/cytologically confirmed lung adenocarcinoma
* Documented ALK-rearrangement mutation positive (assessed by a local laboratory)
* ECOG PS 0-1
* Patients must be treatment-naive for NSCLC and eligible to receive treatment with Lorlatinb.
* Measurable disease, as defined by RECIST v1.1
* Hematology, liver and kidney function are adequate for neoadjuvant therapy.
* Cardiopulmonary function suitable for surgical treatment (ECG, echocardiography, pulmonary function or blood gas analysis).
* Male participants must be willing to use acceptable methods of contraception.
* Female participants of childbearing potential must agree to use acceptable methods of contraception.
* Ability to provide written informed consent.

Exclusion Criteria:

* Mixed squamous cell carcinoma, large cell carcinoma, small cell lung cancer.
* Prior treatment with any systemic anti-cancer therapy for locally advanced NSCLC
* Non-resectable stage IB, II, IIIA or selected IIIB NSCLC evaluated by thoracic surgeons.
* Unable to tolerate curative surgery per anaesthesiologist evaluation.History of organ transplant.
* Pregnant or lactating, or intending to become pregnant during the study
* Evidence of any severe or uncontrolled systemic disease, including uncontrolled hypertension and active bleeding, that the investigator considers to be detrimental to patient participation in the study or to adherence to the protocol.
* Past medical history of Interstitial lung disease (ILD), drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD.
* A clear past history of neurological or psychiatric disorders, including epilepsy or dementia;
* Judgement by investigator that the subject should not participate in the study if the subject is unlikely to comply with the study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response (pCR) Rate | Within 1 month after surgery
  Pathologic complete response (pCR) rate is defined as the percentage of participants with no residual viable tumor in lung primary or lymph nodes as evaluated by systematic pathological review of surgical specimens.

SECONDARY OUTCOMES:
Objective response rate | Within 1 month after surgery
  Preoperative radiological evaluation (as assessed by the investigator according to RECIST v1.1) of the number of complete or partial responses as a proportion of the population in the cohort.
Major Pathologic Response (MPR) Rate | Within 1 month after surgery
  Major pathologic response (MPR) rate is defined as the percentage of participants with less than or equal to 10% of residual viable tumor in lung primary or lymph nodes as evaluated by systematic pathological review of surgical specimens. Viable tumors in situ carcinoma should not be included in MPR calculation.
Rate of lymph node downstaging | within 3 days after the last CT scan before surgery perfomed
  It is defined as the proportion of patients who have completed the neoadjuvant lorlatinib treatment before surgery and have achieved a N stage downing of the tumor as confirmed by CT evaluation after 6 weeks in all patients who have completed the treatment
The delay of operation | The 3rd day of post-operation
  the proportion of patients who have unanticipated delays to surgery >6 weeks after completion of neoadjuvant treatment
The completion rate of operation | The 3rd day of post-operation
  the proportion of patients who have completed the surgery after neoadjuvant lorlatinib treatment
Incidence of Adverse Events | up to 1 month post surgery
  AE captured by CTCAE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Fan F Yang, M.D., Study Chair — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shaw AT, Felip E, Bauer TM, Besse B, Navarro A, Postel-Vinay S, Gainor JF, Johnson M, Dietrich J, James LP, Clancy JS, Chen J, Martini JF, Abbattista A, Solomon BJ. Lorlatinib in non-small-cell lung cancer with ALK or ROS1 rearrangement: an international, multicentre, open-label, single-arm first-in-man phase 1 trial. Lancet Oncol. 2017 Dec;18(12):1590-1599. doi: 10.1016/S1470-2045(17)30680-0. Epub 2017 Oct 23. PMID 29074098
- See also: Phase 1 trial of Lorlatinib for ALK/ROS1 NSCLC patients. — https://www.cancer.org/cancer/lung-cancer/about/key-statistics.html

DOCUMENTS (1):
  • Study Protocol (2024-09-12): https://cdn.clinicaltrials.gov/large-docs/84/NCT06682884/Prot_000.pdf